CLINICAL TRIAL: NCT01028625
Title: Treatment of Functional Impairment in Patients With Heart Failure and Comorbid Depression
Brief Title: Depression and Self-care in Heart Failure
Acronym: DASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201013037; 1R01HL091918 (NIH)
Record Dates: First submitted 2009-12-04; First posted 2009-12-09 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Heart Failure; Depression
Keywords: Heart failure; Depression; Self Care; Cognitive behavior therapy
MeSH Terms: conditions — Heart Failure; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavior Therapy (Active Comparator)
  Interventions: Behavioral: Cognitive Behavior Therapy; Other: Heart Failure Self-care Education
- Usual Care (Other): Participants who are randomly assigned to usual care will receive whatever treatment (if any) for depression their own physician may prescribe. In most cases, treatment (if any is provided) is likely to consist of a serotonin reuptake inhibitor (SSRI) antidepressant such as sertraline or citalopram.
  Interventions: Other: Heart Failure Self-care Education

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — CBT utilizes a variety of strategies and techniques to modify cognitions and behaviors that contribute to depression such as behavioral activation; identifying and challenging distressing thoughts, beliefs, and attitudes; and systematic problem-solving. In this trial, CBT will be integrated with an intervention aimed at improving heart failure self-care, and with attention to primary caregiver stress. The CBT sessions will usually last about 50 minutes and will be scheduled weekly for up to 6 months, with additional maintenance contacts after that. The frequency of sessions will be tapered prior to 6 months if the participant meets the study criteria for depression remission and has acquired relapse-prevention skills.
  Other Names: CBT
  Arms: Cognitive Behavior Therapy
Other: Heart Failure Self-care Education — Participants in both arms will receive heart failure educational material from the Heart Failure Society of America. In addition, a RN will review educational material with participants during baseline visit and with 3 weekly follow up phone calls.
  Other Names: HFE

SUMMARY:
The purpose of the study is to test whether Cognitive Behavior Therapy (CBT) plus heart failure self-care education is superior to "usual care" for depression.

DETAILED DESCRIPTION:
Comorbid depression is common in heart failure, but little is known about how to treat it. This randomized, controlled, efficacy trial will compare cognitive behavior therapy (CBT) to usual care (UC) for depression in heart failure. CBT will be integrated with an intervention to improve heart failure self-care, because depression and inadequate self-care are thought to be interrelated problems. It will also be integrated with clinical attention to primary caregiver stress. Basic heart failure education will be provided to all participants.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association Class I, II, or III Heart Failure (Clinically diagnosed at least 3 months ago)
* Meets the DSM-IV criteria for a current major depressive episode, or for current minor depression with a past history of at least one major depressive episode.
* PHQ-9 score of 10 or greater plus 2 or 3 on question 1 or 2 over the last 2 weeks including today

Exclusion Criteria:

* Less than 30 years old
* Current ETOH / drug abuse
* Bipolar disorder, schizophrenia, or other psychotic disorder
* Communication barrier
* Dementia
* Currently in competing research protocol
* High risk for suicide
* Insurmountable logistical barriers to laboratory assessment visits
* Major mobility-limiting physical disability
* Poor 1 year prognosis not r/t heart failure
* Hospitalized for heart failure or acute coronary syndrome in last month
* Initiated antidepressant therapy in the past 4 weeks
* Current non-study psychotherapy for depression or other psychiatric problem

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2010-01; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
BDI-II score at 6 months | Baseline, 3 months, 6 months, 9 months , 12 months

SECONDARY OUTCOMES:
Self-care of Heart Failure Index | Baseline, 3 months, 6 months, 9 months, 12 months
Beck Anxiety Inventory | Baseline, 3 months, 6 months, 9 months, 12 months
Medical outcomes study SF-12 | Baseline, 3 months, 6 months, 9 months, 12 months
PROMIS Physical Functioning Scale | Baseline, 6 months
Kansas City Cardiomyopathy Questionnaires | Baseline, 3 months, 6 months, 9 months, 12 months
6 Minute Walk Test | Baseline, 6 months
Depression Interview and Structured Hamilton (DISH) | Baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E. Freedland, Ph.D., Principal Investigator — Washington University School of Medicine Behavioral Medicine Center
Locations (1):
- Washington University School of Medicine Behavioral Medicine Center, St Louis, Missouri, United States

REFERENCES:
- [Derived] Smagula SF, Freedland KE, Steinmeyer BC, Wallace MJ, Carney RM, Rich MW. Moderators of Response to Cognitive Behavior Therapy for Major Depression in Patients With Heart Failure. Psychosom Med. 2019 Jul/Aug;81(6):506-512. doi: 10.1097/PSY.0000000000000712. PMID 31083052
- [Derived] Freedland KE, Steinmeyer BC, Carney RM, Rubin EH, Rich MW. Use of the PROMIS(R) Depression scale and the Beck Depression Inventory in patients with heart failure. Health Psychol. 2019 May;38(5):369-375. doi: 10.1037/hea0000682. PMID 31045419
- [Derived] Freedland KE, Carney RM, Rich MW, Steinmeyer BC, Rubin EH. Cognitive Behavior Therapy for Depression and Self-Care in Heart Failure Patients: A Randomized Clinical Trial. JAMA Intern Med. 2015 Nov;175(11):1773-82. doi: 10.1001/jamainternmed.2015.5220. PMID 26414759